CLINICAL TRIAL: NCT04846725
Title: Predictors of Attempted Inferior Vena Cava Filters Retrieval.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN372021/CHUSTE
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Venous Thromboembolic Disease
Keywords: Inferior vena cava filter; inferior vena cava filter retrieval; inferior vena cava filter complications; deep vein thrombosis (DVT); pulmonary embolism; venous thromboembolism event (VTE)
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrievable Inferior Vena Cava Filters (IVCF): The population study includes patients with a Retrievable Inferior Vena Cava Filters (IVCF) inserted between April 2012 and November 2019. Follow up data is collected up to July 2020.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Collect in medical records :
  * Filter's retrieval rate
  * Complications of vena cava filters
  * Predictive factors of attempted inferior vena cava filters retrieval: age, the distance between the patient's home and the hospital, the indication or not given by the therapeutic medicine department, patients referred by external structures, patients whose filter was installed during the medical on-call period, the absence of a written request for filter placement, the presence of active neoplasia at the time of filter placement, a peri-surgical context.

SUMMARY:
The InferiorVena Cava (IVC) with filters has been recommended when there is a contraindication or a failure of anticoagulation. Due to the side effects related to the filters, it is recommended to remove them as soon as possible. It's a retrospective study in a French hospital to evaluate the retrieval rate and predictors of filter removal.

All the data of consecutive patients who had a retrievable InferiorVena Cava Filter (IVCF) inserted in the investigator center between April 2012 and November 2019 are included.

ELIGIBILITY:
Inclusion Criteria:

* patients who had a cave filter placement at Saint-Etienne Hospital between april 2012 and november 2019.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had a cave filter placement at Saint-Etienne Hospital between april 2012 and november 2019 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Filter's retrieval rate (%) | Month: 2
  Collect in medical records.

SECONDARY OUTCOMES:
Predictive factors of attempted inferior vena cava filters retrieval | Month: 2
  Collect in medical records.
Adverse event of vena cava filters | Month: 2
  Collect in medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Grange, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No